CLINICAL TRIAL: NCT01776294
Title: Prevalence of Prehypertension Among Medical Students and Association With Cardiovascular Risk Factors
Brief Title: Prehypertension Among Medical Students in Visakhapatnam and Association With Cardiovascular Risk Factors
Status: Completed | Type: Observational
Sponsor: Andhra Medical College (Other Government)
Responsible Party: Principal Investigator, Ravi Venkatachelam Chitrapu, Associate Professor, Andhra Medical College
Other Study IDs: 04AMCRVCTZM12
Record Dates: First submitted 2012-12-25; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Prehypertension; Cardiovascular Risk Factors
Keywords: Prehypertension; Prevalence; Cardiovascular Risk Factors
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- prehypertensives: students will be classified as prehypertensives as per the JNC-7 (Joint National Commission) guidelines based on their Blood Pressure measurement
- normotensives: students will be classed as normotensives based on their BP measurement as per JNC-7 guidelines (systolic <120 AND diastolic <80)

SUMMARY:
Student Investigator = Thakkallapalli Zeeshan Muzahid. The study aims to assess the prevalence of prehypertension among medical students of Andhra Medical College, Visakhapatnam, India and its association with other cardiovascular risk factors - overweight /obesity, diabetes, lipid profile.

DETAILED DESCRIPTION:
275 medical students will be studied and a history taken and examination done with special emphasis on recording of Blood Pressure, measurement of height and weight (& Body Mass Index) and Waist Circumference in all. Glucose Tolerance Test and Fasting Lipid profile will be measured in a random selection of 30 prehypertensives and 30 normotensives.

ELIGIBILITY:
Inclusion Criteria:

* Medical Students studying MBBS (Bachelor of Medicine & Bachelor of Surgery) in Andhra Medical College
* clinically healthy
* consent to participate in the study

Exclusion Criteria:

* known cardiovascular disease
* known hypertension
* using antihypertensive or other cardiovascular drugs
* using any drugs that can affect BP, weight, Blood sugar

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Graduate Medical Students
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
prevalence of prehypertension among graduate medical students | two weeks
  the point prevalence of prehypertension at the time of survey will be estimated - as the students were examined over two weeks

SECONDARY OUTCOMES:
correlation between blood pressure (Prehypertension) and BMI (obesity), Blood glucose, LDL level (dyslipidemia) | two weeks
  correlation of prehypertension with Body Mass Index, Waist Circumference (for overweight /obesity) smoking and blood glucose levels and lipid profile - time frame was given as two weeks as that was the period during which the students were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Thakkallapalli Zeeshan Muzahid, MBBS, Principal Investigator — Andhra Medical College
Locations (1):
- Andhra Medical College, Visakhapatnam, Andhra Pradesh, India